CLINICAL TRIAL: NCT05466825
Title: Predicting Cardiovascular Risk by Geographical Region and Sex Using Classical Cardiovascular Risk Factors
Brief Title: The Global Cardiovascular Risk Consortium
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Blankenberg, Prof. Dr. med., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: GCVRC001
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: All-cause Mortality; Cardiovascular Disease
Keywords: Cardiovascular Disease; Cardiovascular Risk Factors; Risk Factor Modification; Global; Lifetime Gain
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Global Cardiovascular Risk Consortium (GCVRC) brings together harmonized individual-level data from over 2 million individuals across 133 cohorts, 39 countries, and 6 continents, with recruitment ongoing. The GCVRC examines the impact of classical cardiovascular risk factors-such as body mass index, systolic blood pressure, non-high-density lipoprotein cholesterol, current smoking, and diabetes-on cardiovascular disease (CVD) and death from any cause worldwide.

DETAILED DESCRIPTION:
A small number of modifiable risk factors may account for a significant proportion of cardiovascular disease (CVD) risk. However, the CVD burden attributable to classical risk factors depends on the populations studied and the methodologies used.

The Global Cardiovascular Risk Consortium (GCVRC) is an international collaboration that continuously includes cohort studies from around the world to improve cardiovascular risk prediction. The GCVRC uses extensively harmonized individual-level data from currently more than 2 Mio individuals from 133 cohorts, 39 countries and 6 continents categorized in 8 geographical regions (based on a modification of WHO and United Nations definitions) - North America, Latin America, Sub-Saharan Africa, North Africa and the Middle East, Western Europe, Eastern Europe and Russia, Asia, and Oceania.

The consortium has a special focus on classical, potentially modifiable cardiovascular risk factors: Body-mass index, systolic blood pressure, non-high-density lipoprotein cholesterol, current smoking, and diabetes. Key research questions include examining the impact of these factors on major outcomes by geographical region and sex, as well as estimating associated lifetime risk and the potential lifetime difference when modifying these risk factors.

This work is critical for developing regionally tailored CVD prevention and treatment strategies, identifying residual risk, and improving global cardiovascular health. Based on GCVRC data, a landmark paper on the effect of classical risk factors on new-onset CVD and all-cause mortality was published in the New England Journal of Medicine in 2023 (https://doi.org/10.1056/nejmoa2206916).

ELIGIBILITY:
Inclusion Criteria:

Population-based individual-level data with available information on the classical cardiovascular risk factors including body-mass index, systolic blood pressure, non-high-density lipoprotein cholesterol, current smoking, and diabetes, as well as the outcomes of interest.

Exclusion Criteria:

* Participants with age below 18 years
* No information on the outcome of interest
* No information on the exposure of interest (CVD risk factors)
* History of CVD at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The GCVRC uses harmonized individual-level data from currently more than 2 Mio individuals from 133 cohorts, 39 countries and 6 continents, categorized in 8 geographical regions - North America, Latin America, Sub-Saharan Africa, North Africa and the Middle East, Western Europe, Eastern Europe and Russia, Asia, and Oceania.
  The database provides information on cardiovascular risk factors, including body-mass index, systolic blood pressure, non-high-density lipoprotein cholesterol, current smoking, and diabetes, as well as data on major outcomes.
Sampling Method: Probability Sample
Enrollment: 2500000 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease (CVD) | Median follow-up of 7-10 years
  Event rates of CVD and CVD subtypes: First fatal or non-fatal myocardial infarction, unstable angina, coronary revascularization, ischemic or hemorrhagic stroke, and cardiovascular or unclassifiable death. The type of outcome measurement varies across cohorts. CVD cases and subtypes are assessed by questionnaire information, national hospital discharge registry data, causes of death registry data or central death registries depending on the study protocol of the respective cohort studies.
All-cause mortality (ACM) | Median follow-up of 7-10 years
  Number of deaths from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Stefan Blankenberg, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Cardiovascular Risk Consortium; Magnussen C, Ojeda FM, Leong DP, Alegre-Diaz J, Amouyel P, Aviles-Santa L, De Bacquer D, Ballantyne CM, Bernabe-Ortiz A, Bobak M, Brenner H, Carrillo-Larco RM, de Lemos J, Dobson A, Dorr M, Donfrancesco C, Drygas W, Dullaart RP, Engstrom G, Ferrario MM, Ferrieres J, de Gaetano G, Goldbourt U, Gonzalez C, Grassi G, Hodge AM, Hveem K, Iacoviello L, Ikram MK, Irazola V, Jobe M, Jousilahti P, Kaleebu P, Kavousi M, Kee F, Khalili D, Koenig W, Kontsevaya A, Kuulasmaa K, Lackner KJ, Leistner DM, Lind L, Linneberg A, Lorenz T, Lyngbakken MN, Malekzadeh R, Malyutina S, Mathiesen EB, Melander O, Metspalu A, Miranda JJ, Moitry M, Mugisha J, Nalini M, Nambi V, Ninomiya T, Oppermann K, d'Orsi E, Pajak A, Palmieri L, Panagiotakos D, Perianayagam A, Peters A, Poustchi H, Prentice AM, Prescott E, Riserus U, Salomaa V, Sans S, Sakata S, Schottker B, Schutte AE, Sepanlou SG, Sharma SK, Shaw JE, Simons LA, Soderberg S, Tamosiunas A, Thorand B, Tunstall-Pedoe H, Twerenbold R, Vanuzzo D, Veronesi G, Waibel J, Wannamethee SG, Watanabe M, Wild PS, Yao Y, Zeng Y, Ziegler A, Blankenberg S. Global Effect of Modifiable Risk Factors on Cardiovascular Disease and Mortality. N Engl J Med. 2023 Oct 5;389(14):1273-1285. doi: 10.1056/NEJMoa2206916. Epub 2023 Aug 26. PMID 37632466
- [Derived] Global Cardiovascular Risk Consortium; Magnussen C, Alegre-Diaz J, Al-Nasser LA, Amouyel P, Aviles-Santa L, Bakker SJL, Ballantyne CM, Bernabe-Ortiz A, Bobak M, Boffetta P, Brenner H, Brunstrom M, Can G, Carrillo-Larco RM, Checkley W, Dallongeville J, De Bacquer D, de Gaetano G, de Lemos JA, di Carluccio E, Dobson A, Donfrancesco C, Dorr M, d'Orsi E, Drygas W, Dullaart RPF, Engstrom G, Ferrario MM, Ferrieres J, Figtree GA, Gaye B, Ghayour-Mobarhan M, Goldbourt U, Gonzalez C, Gossling A, Grassi G, Gupta PC, He J, Hodge AM, Hozawa A, Hveem K, Iacoviello L, Ikram MK, Inoue M, Irazola V, Jobe M, Jousilahti P, Kaleebu P, Kavousi M, Kee F, Khalili D, Klotsche J, Koenig W, Kontsevaya A, Kowlessur S, Kuri-Morales P, Kuulasmaa K, Kweon SS, Lackner KJ, Landmesser U, Leistner DM, Leiva Sisnieguez CE, Leong D, Lind L, Linneberg A, Lorenz T, Lyngbakken MN, Malekzadeh R, Malyutina S, Mathiesen EB, McElduff P, Melander O, Metspalu A, Miranda JJ, Moitry M, Mugisha J, Munzinger J, Nalini M, Nambi V, Nilsson PM, Ninomiya T, Omland T, Ong SK, Oppermann K, Pajak A, Palmieri L, Panagiotakos D, Park SK, Pednekar MS, Perianayagam A, Peters A, Poustchi H, Prabhakaran D, Prentice AM, Prescott E, Quyyumi A, Riserus U, Sakata S, Salazar M, Salomaa V, Sans S, Sattler ELP, Schottker B, Schutte AE, Sepanlou SG, Sharma SK, Shaw J, Simons LA, Soderberg S, Tamosiunas A, Tapia-Conyer R, Thorand B, Tunstall-Pedoe H, Tuomilehto J, Twerenbold R, Vanuzzo D, Veronesi G, Wannamethee SG, Watanabe M, Weimann J, Wild PS, Yao Y, Zeng Y, Ziegler A, Ojeda FM, Blankenberg S; The Global Cardiovascular Risk Consortium. Global Effect of Cardiovascular Risk Factors on Lifetime Estimates. N Engl J Med. 2025 Jul 10;393(2):125-138. doi: 10.1056/NEJMoa2415879. Epub 2025 Mar 30. PMID 40162648